CLINICAL TRIAL: NCT06765135
Title: Point of Care Respiratory Pathogen Testing for Antibiotic Stewardship in Primary Care
Acronym: PROTECT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Lauren Dutcher, Assistant Professor of Medicine, University of Pennsylvania
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 856091
Record Dates: First submitted 2024-12-11; First posted 2025-01-09 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-12

CONDITIONS: Upper Respiratory Infection
Keywords: upper respiratory infections; primary care clinics; point of care testing; antibiotic stewardship
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Focus Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clinicians/practice staff (Other): Clinicians will be the target for the intervention that will include provision of the POC RPP (Point of Care Respiratory Pathogen Panel) test as well as clinical guidance on use and interpretation. Clinicians will also be included in focus groups and surveys, and other administrative practice staff will also be included in focus groups. All clinicians/staff practicing at one of the included practices will be eligible for inclusion
  Interventions: Behavioral: Clinician Survey; Behavioral: Focus Group; Diagnostic Test: Biofire Spotfire Respiratory (R) panel
- Patients (Other): All adult patients (age >=18 years) at one of the included primary care practices seen for an upper respiratory infection or symptom will be included in the primary study analysis, as identified by ICD-10 code (from baseline and intervention periods). Patients with ICD-10 codes for other bacterial infections at the same encounter will be excluded (e.g., skin and soft tissue infection) from the analysis. During the intervention period, adult patients with symptoms potentially suggestive of an upper respiratory infection will be eligible for use of the POC RPP test.
  Interventions: Diagnostic Test: Biofire Spotfire Respiratory (R) panel; Behavioral: Patient Survey

INTERVENTIONS:
Behavioral: Clinician Survey — At the conclusion of the intervention period, practice stakeholders, including survey providers and practice managers in the intervention sites will be surveyed to identify their degree of satisfaction with the intervention and suggestions for improvement.
  Arms: Clinicians/practice staff
Behavioral: Focus Group — Prior to installing the device in each primary care practice, trained moderators will conduct focus groups with clinicians and practice staff to to elicit provider perceptions of POC testing for respiratory pathogens, including feasibility and acceptability of integration of testing into routine workflows.
  Arms: Clinicians/practice staff
Diagnostic Test: Biofire Spotfire Respiratory (R) panel — Eligible patients will be offered testing with the BioFire Spotfire Respiratory (R) Panel, which is an FDA-cleared, CLIA waived test. This is a multiplexed polymerase chain reaction (PCR) test intended for use with the BioFire Spotfire System for the simultaneous, qualitative detection and identification of multiple respiratory viral and bacterial nucleic acids in nasopharyngeal (NP) swab specimens obtained from individuals with signs and symptoms of respiratory tract infection, including COVID-19. This testing will be made available in participating practices along with clinical guidance about use and interpretation. Clinicians will administer the tests to patients who agree to be tested. Results will be shared with patients, who can discuss the results with their clinicians. Clinicians can use the test results to guide their treatment decisions.
Behavioral: Patient Survey — During the intervention period, patients who undergo POC RPP testing will be surveyed soon after their visit to elicit their opinions about the test.
  Arms: Patients

SUMMARY:
The goal of this study is to understand the use of point of care (POC) testing devices in primary care offices to help clinicians diagnose and appropriately treat patients who have symptoms of upper respiratory infections (URIs).

The study will use the BIOFIRE® SPOTFIRE® Respiratory (R) Panel testing device, which is FDA-cleared and CLIA-Waived. This panel can identify up to 15 different viruses and bacteria that can cause URIs.

These POC devices will be installed in primary care clinics within the University of Pennsylvania Health System. Patients who come to the clinic with cold-like symptoms (runny nose, cough) will be offered the test. If the patient agrees to the test, their clinician will use a swab to take a small sample of fluid from their nose. This swab will then be tested within the POC device and results will be available within 15 minutes.

The results of this sample will be shared with the patient, and their clinician can use the results to help decide the most appropriate medical treatment for the patient.

Patients who agree to take the test will be asked to answer a short survey about the test and their experience. Clinicians will also be surveyed to share their thoughts with using the test in their clinics. Focus groups of practice staff and clinicians will also be conducted to understand any potential challenges for using this test in practice.

Results from the tests and the surveys will help researchers understand the value of the test to support antibiotic stewardship efforts in primary care clinic settings.

DETAILED DESCRIPTION:
Point of care (POC) testing for respiratory viral pathogens has been proposed as a potential tool for use in antibiotic stewardship in primary care, particularly with reducing diagnostic uncertainty and supporting providers in communication about upper respiratory symptom etiology. However, there are limited data to support their widespread use. The research team propose to conduct a study that seeks to understand the role of POC respiratory pathogen testing on antibiotic prescribing in primary care practices. The research team plan to use qualitative methods, including focus groups and surveys of primary care clinicians to understand provider perceptions of POC respiratory pathogen testing (part 1). The research team will then perform a pragmatic, stepped-wedge, cluster randomized trial in 4-8 primary care practices to study the impact of implementation of the POC respiratory pathogen testing, using the Spotfire R panel, on antibiotic prescribing (part 2). The results from part 1 of the study will be used to optimize implementation in part 2 of the study. The research team will also assess several secondary outcomes in part 2, including antiviral prescribing, healthcare utilization, and patient and provider perceptions of the use of POC respiratory pathogen testing.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* Symptoms of an upper respiratory infection to include: cough, rhinorrhea, nasal congestion, fever, sore throat, ear pain/fullness, sinus pain

Exclusion Criteria:

* Age < 18 years of age
* No relevant upper respiratory symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Antibiotic prescription at index visit | From participant enrollment to end of index visit
  Proportion of patients with an antibiotic prescribed at the index visit

SECONDARY OUTCOMES:
Provider attitudes and perceptions toward point of care respiratory pathogen testing | Two months following completion of study intervention
  Attitudes and perceptions reported by providers on the "PROTECT Clinician Survey" instrument
Patient attitudes and perceptions toward point of care respiratory pathogen testing | From participant enrollment to two weeks after index visit
  Attitudes and perceptions reported by patients on the "PROTECT Patient Survey" instrument
Antiviral prescription at index visit | From participant enrollment to end of index visit
  Proportion of patients with an antiviral prescribed at the index visit
Antibiotic prescription at index visit for specific subgroups, including patients with specific diagnoses (sinusitis, acute bronchitis, acute pharyngitis) and patients with ICD-10 codes for diagnoses for which an antibiotic is typically not warranted | From participant enrollment to end of index visit
  Proportion of patients with an antibiotic prescribed at the index visit within specific subgroups, including patients with sinusitis, acute bronchitis, acute pharyngitis, and patients with diagnoses for which an antibiotic is not typically warranted
Healthcare utilization, to include: 1. Follow up visits within 14 days after the index visit 2. Follow up telephone calls and messages within 14 days after the index visit 3. Antibiotic or antiviral prescriptions within 14 days after the index visit | From participant enrollment to 14 days after index visit
  Proportion of patients with 1) follow up visits; 2) follow up telephone calls or messages; 3) antibiotic prescribed; 4) antiviral prescribed within 14 days following the index visit
Test utilization, to include use of Spotfire R panel | From participant enrollment to 14 days after index visit
  Proportion of patients who underwent POC RPP (Point of Care Respiratory Pathogen Panel) testing at the index visit
Test utilization, to include laboratory-based respiratory pathogen testing | From participant enrollment to 14 days after index visit
  Proportion of patients who underwent testing for respiratory viruses using laboratory-based testing at the index visit
Test utilization, to include Group A streptococcal testing | From participant enrollment to 14 days after index visit
  Proportion of patients who underwent testing for group A streptococcus at the index visit
Test utilization, to include chest imaging | From participant enrollment to 14 days after index visit
  Proportion of patients ordered for chest imaging at the index visit

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania Primary Care Practice, Philadelphia, Pennsylvania, United States